CLINICAL TRIAL: NCT05628220
Title: Evaluation and Countermeasures of Motion Sickness by Virtual Reality Desensitization Protocol
Brief Title: Motion Sickness Desensitization Using VR
Acronym: SENSORIEL1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-083
Record Dates: First submitted 2022-09-08; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-08

CONDITIONS: Motion Sickness
Keywords: vestibular system; posture; anxiety; nausea; motion sickness; visually induced motion sickness
MeSH Terms: conditions — Motion Sickness; Anxiety Disorders; Nausea | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: one cohort of patients suffering from motion sickness
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort of motion sickness (Other): one group of patient
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: physiotherapy — rehabilitation through using session of virtual reality desensitization

SUMMARY:
Evaluation of a virtual reality desensitization protocol on subjects with severe motion sickness and study of the role of the emotional component on the effectiveness of the therapy.

DETAILED DESCRIPTION:
Motion sickness is a well-known syndrome, particularly at risk in children, with a maximum around the age of 12. All people are sensitive to motion sickness in childhood, probably related to the maturation of certain cognitive functions of a spatial nature, namely the perception of oneself and one's movements in one's environment. These symptoms regress with age for a part of the population but a large number of people will remain sensitive to certain conditions of displacement and generate symptoms that can be extremely disabling and handicapping in everyday life, particularly for professional activities. For example, some people can no longer use their car, some can no longer take the boat for professional activities in restrictive and/or extreme environments (sailors, scientists, workers, etc.). Behavioral, respiratory or medicinal therapies remain partially effective due to the lack of sufficient knowledge on the physiopathology of this syndrome classified in the field of sensory disorders. Very recently, techniques of sensory desensitization by visual stimulation have appeared, either optokinetic or in virtual reality mimicking the environment that causes this syndrome. This therapeutic approach seems to give empirically good results but only one study has shown it with optokinetic stimulation but it is to be evaluated for virtual reality.

The main objective of the study is therefore to evaluate the effectiveness of a sensory conflict protocol generated in virtual reality to reduce the severity of motion sickness. Each subject being his own control. An observational study was then designed to quantify the effectiveness of this technique carried out in a current way by the physiotherapists in the form of questionnaires supplemented by a posturographic evaluation of the sensory profile of the subjects. If the effectiveness is proven, this desensitization protocol could be optimized and more widely distributed. Furthermore, the analysis of the visuo-dependence variable (from the sensory profile) will indicate whether the use of a visual stimulus by virtual reality alone is sufficient or should be combined or compared with desensitization of other sensory modalities. The use of galvanic vestibular stimulation for the rehabilitation of vestibular pathologies or training programs based on the resolution of sensory conflicts could be envisaged in the future.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from motion sickness inducing a functional disability requiring a change in the mode of travel, or suffering from motion sickness disabling to exercise a leisure or professional activity involving a mode of locomotion.

Exclusion Criteria:

* Pregnant woman
* History of severe ENT or ophthalmologic pathologies.
* Chronic treatment with an anticholinergic or anti-histamine medication.
* Participating in another biomedical research protocol during the same period
* Person under guardianship or curatorship

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
motion sickness severity | day 0 (day before the first session of rehabilitation)
  simulator sickness questionnaire (0-64)
motion sickness severity | day 30 (day after the end of rehabilitation)
  simulator sickness questionnaire (0-64)

SECONDARY OUTCOMES:
Emotion | day 0 (day before the first session of rehabilitation)
  The State-Trait Anxiety Questionnaire (0-80)
Emotion | day 30 (day after the end of rehabilitation)
  The State-Trait Anxiety Questionnaire (0-80)
Posture | day 0 (day before the first session of rehabilitation)
  postural measurement (gravity center ellipse)
Posture | day 30 (day after the end of rehabilitation)
  postural measurement (gravity center ellipse)

CONTACTS AND LOCATIONS:
Overall Officials: stephane BESNARD, Md,PhD, Principal Investigator — University Hospital, Caen
Locations (2):
- France (2):
  - Caen University Hospital, Caen
  - Frédéric Xavier, Vitrolles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: topical team motion sickness — https://gdrvertige.com/